CLINICAL TRIAL: NCT03207659
Title: Dusting vs Basketing in RIRS: a Single-center Prospective Randomised Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guohua Zeng (Other)
Responsible Party: Sponsor-Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dusting vs Basketing in RIRS
Record Dates: First submitted 2017-06-24; First posted 2017-07-05 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Urolithiasis
Keywords: RIRS; Renal stones; Efficacy; Safety
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis | interventions — Dust

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dusting (Experimental): small stones will be left to pass spontaneously.
  Interventions: Procedure: Dusting in RIRS
- Basketing (Experimental): stones will be actively extracted.
  Interventions: Procedure: Basketing in RIRS

INTERVENTIONS:
Procedure: Basketing in RIRS — Treament of renal stones by fragmentation of stone under direct vision through a flexible ureteroscope and then actively extracting them using a basket
  Arms: Basketing
Procedure: Dusting in RIRS — Treament of renal stones by dusting the stone under direct vision through a scope and then leaving them to pass spontaneously
  Arms: Dusting

SUMMARY:
The investigator aims to perform a prospective and randomized controlled trial comparing the safety and efficacy of active basket extraction of fragments and stone dusting during the RIRS.

DETAILED DESCRIPTION:
RIRS has been widely adopted and used by urologists worldwide in the management of renal stones due to less invasiveness and efficacy, especially in small to moderate-sized renal stones. RIRS has several advantages over SWL for stones less than 2 cm diameter. Most importantly, removing the stone in one session without the need for other treatment modalities.

Furthermore, the application of RIRS has expanded to larger stones reaching up to 35 mm in some cases,in spite of not being the first line therapy for the larger stones. RIRS has advantages over the PCNL especially concerning complications. Namely lower or no bleeding events and the less invasiveness of RIRS.

Options for the treatment of intrarenal stones include fragmenting the stone then extracting large fragments using a basket or dusting the stone into very small fragments then leaving the (dust) to pass spontaneously.

The idea of dusting in RIRS emerges as a counterpart of the originally taught fragmentation and basketing of the stones. Aiming to reduce multiple entries and exits for the renal system and ultimately not requiring UAS or baskets during the surgery. Thus theoretically decreasing operative time and costs with the same SFRs, In addition to minimizing the risk of ureteral injury .

So there is a debate amongst surgeons whether to laser the stone to dust or fragment and retrieve intra-renal fragments. EAU guidelines on the surgical management of urolithiasis stated that dusting strategies should be limited to the treatment of large renal stones. Without clearly differentiating between dusting or fragmentation and basketing. Cho et al; favored fragmentation technique especially for large renal stones because the dust in dusting technique may affect visualization and obscure small stone fragments. But this was an opinion and not built on a direct comparative study.

Until now, there is no consensus on how to achieve optimal stone clearance once the primary stone is fragmented with lithotripsy. And to date, no prospective randomized study has addressed the practice of active extraction vs. spontaneous passage

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be a suitable operative candidate for RIRS
2. Age ≥18 years
3. Normal renal function
4. ASA score Ⅰ and Ⅱ
5. Single renal stone ≤20mm or multiple stones the conglomerate diameter (additive maximal diameter of all stones on axial imaging of computed tomography) up to 20 mm

Exclusion Criteria:

1. Pregnant subjects
2. Uncorrected coagulopathy and active urinary tract infection (UTI)
3. prior ipsilateral endourological procedure history, such as RIRS, PCNL, URS and URL
4. Patients who underwent transplant or urinary diversion.
5. Congenital abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Stone free rate (SFR) | 4-6 weeks after surgery
  To assess for stone-free rate using K.U.B. (kidney-ureter-bladder) plain radiograph and renal ultrasound. If there is a discrepancy in follow up imaging between the presence of residual stones or fragments between the KUB and renal ultrasound, the KUB will be considered the reference standard for small fragments less than 4mm unless the stone composition is uric acid. If fragments 5 mm or larger exist or uric acid it will be up to the discretion of the surgeon to order a CT to better delineate the presence of residual stones and their impact on the clinical management of that patient.

SECONDARY OUTCOMES:
Operating time | intraoperatively
  from starting fragmentation to placement of stent (DJ stent or ureteral stent) unless no stent is needed
Complication rates | intraoperatively or 48h postoperatively
  Complication such as fever, pain, urosepsis etc.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D & MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No